CLINICAL TRIAL: NCT02003612
Title: An Analysis of Historical Data on Hematological Remission and Survival Among Adult Patients With Relapsed / Refractory B-Precursor Acute Lymphoblastic Leukemia
Brief Title: Historical Data Analysis of Hematological Remission and Survival in Adults With R/R Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20120310
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All subjects: All subjects
  Interventions: Other: Not applicable - observational study

INTERVENTIONS:
Other: Not applicable - observational study — No intervention exists as this is a retrospective observational study

SUMMARY:
A retrospective analysis of historical data looking at hematological remission and survival in adult relapsed / refractory B-precursor acute lymphoblastic leukemia patients.

DETAILED DESCRIPTION:
A retrospective observational study reviewing historical survival data (hematological remission and survival) for adult patients who have either relapsed or refractory B-precursor acute lymphoblastic leukemia. Data are aggregated across multiple countries and study sites in the EU and US

ELIGIBILITY:
Inclusion Criteria:

* adult patients with relapsed / refractory B-precursor acute lymphoblastic leukemia
* age 15 or older at time of de novo (initial) diagnosis of acute lymphoblastic leukemia
* initial diagnosis of acute lymphoblastic leukemia in the year 1990 or later
* No CNS involvement at relapse
* No isolated extramedullary relapse
* Other inclusion criteria may apply

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with relapsed / refractory B-precursor acute lymphoblastic leukemia identified in study group databases from multiple sites in EU and US
Sampling Method: Non-Probability Sample
Enrollment: 2373 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2014-01-10 (Actual); Study Completion 2014-04-28 (Actual)

PRIMARY OUTCOMES:
hematological complete remission | Approx 1 year
  To estimate the proportion of patients in hematological complete remission (CR) for R/R Philadelphia chromosome negative (Ph-) B-precursor ALL patients following relapse or salvage treatment, excluding patients with a first remission duration of >12 months in first salvage (ie, patients with late relapse in first salvage)

SECONDARY OUTCOMES:
overall survival | Approx 1 year
  to estimate overall survival for relapsed / refractory philadelphia negative B-precursor acute lymphoblastic leukemia patients following salvage treatment, excluding patients with late relapse in first salvage
duration of complete remission | Approx 1 year
  to estimate the duration of complete remission for philadelphia negative patients following treatment for relapsed / refractory B-precursor acute lymphoblastic leukemia, excluding patients with late relapse in first salvage
proportion of patients receiving allogeneic hematological stem cell transplantation | Approx 1 year
  estimate the proportion of patients receiving allogeneic hematological stem cell transplantation for philadelphia negative patients following treatment for relapsed / refractory B-precursor acute lymphoblastic leukemia excluding those with late relapse in first salvage

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (10):
- United States (2):
  - Research Site, Boston, Massachusetts
  - Research Site, Cleveland, Ohio
- Research Site, Brno, Czechia
- Research Site, Paris, France
- Research Site, Frankfurt am Main, Germany
- Italy (2):
  - Research Site, Bologna
  - Research Site, Venezia
- Research Site, Gliwice, Poland
- Research Site, Badalona, Catalonia, Spain
- Research Site, London, United Kingdom

REFERENCES:
- [Derived] Barlev A, Lin VW, Katz A, Hu K, Cong Z, Barber B. Estimating Long-Term Survival of Adults with Philadelphia Chromosome-Negative Relapsed/Refractory B-Precursor Acute Lymphoblastic Leukemia Treated with Blinatumomab Using Historical Data. Adv Ther. 2017 Jan;34(1):148-155. doi: 10.1007/s12325-016-0447-x. Epub 2016 Nov 21. PMID 27873237
- [Derived] Gokbuget N, Dombret H, Ribera JM, Fielding AK, Advani A, Bassan R, Chia V, Doubek M, Giebel S, Hoelzer D, Ifrah N, Katz A, Kelsh M, Martinelli G, Morgades M, O'Brien S, Rowe JM, Stieglmaier J, Wadleigh M, Kantarjian H. International reference analysis of outcomes in adults with B-precursor Ph-negative relapsed/refractory acute lymphoblastic leukemia. Haematologica. 2016 Dec;101(12):1524-1533. doi: 10.3324/haematol.2016.144311. Epub 2016 Sep 1. PMID 27587380
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com